CLINICAL TRIAL: NCT02215369
Title: Prospective Safety and Effectiveness Study: VenaCure Endovenous Laser Treatment (EVLT) 400 µm Fiber Procedure Kit for Treatment of Incompetent Perforator Veins
Brief Title: SeCure Endovenous Laser Treatment Study
Acronym: SeCure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV-VC300
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VenaCure EVLT 400 µm fiber Procedure Kit (Experimental): Only one limb can be treated and included in this study; however, multiple IPV's within the study limb may be treated. All IPV's treated will be followed according to the study schedule.
  Interventions: Device: VenaCure EVLT 400 µm fiber Procedure Kit

INTERVENTIONS:
Device: VenaCure EVLT 400 µm fiber Procedure Kit — The study intervention will be conducted according to the DFU included with the VenaCure EVLT 400 µm fiber Procedure Kit.

SUMMARY:
The VenaCure EVLT 400 µm Fiber Kit is currently marketed for the treatment of varicose veins. AngioDynamics, Inc., the company that manufacturers the VenaCure device, is sponsoring this study to assess the safety and effectiveness of the VenaCure EndoVenous Laser Treatment (EVLT) 400 µm Fiber Kit for treatment of incompetent perforator veins (IPVs). The VenaCure EVLT 400 µm Fiber Kit has not been previously studied by AngioDynamics for the ablation of IPVs.

DETAILED DESCRIPTION:
This is a single-arm, prospective, multicenter, non-blinded clinical trial. Study data will be summarized and submitted to the FDA in a premarket notification once all treated subjects have completed the 3 month visit. Longer term followup is being performed for publication purposes.

Patients diagnosed with incompetent Perforator Veins (IPV's) and meet all inclusion and none of the exclusion criteria will be eligible for this study.

ELIGIBILITY:
INCLUSION CRITERIA

Patients are required to fulfill all the following criteria to be included in the study:

1. Is ≥ 18 years of age
2. IPV(s) to be treated have an outward flow duration of ≥ 0.5 sec immediately after manual release of manual compression
3. IPV(s) to be treated have a diameter of ≥ 3.5 mm (measured at the level of the fascia) located superior to foot and distal ankle
4. Has been diagnosed with refractory symptomatic disease (CEAP Class 4b to Class 6) attributable to the IPV to be treated
5. Has palpable pedal pulses in the study limb
6. Any pathologic superficial saphenous veins have been previously eliminated and were done so at least more than 30 days prior to the study procedure
7. Is able to ambulate
8. Is able to comprehend and have signed the Informed Consent Form (ICF) to participate in the study
9. Is willing and able to comply with the Clinical Investigation Plan and follow-up schedule

EXCLUSION CRITERIA

Patients will be excluded from participation in the study if they meet any of the following:

1. Has venous insufficiency secondary to venous obstruction proximal to the intended treatment site
2. Has thrombus in the vein segment to be treated
3. Has known peripheral arterial disease
4. Has a BMI calculation (BMI = W / H2 ) ≥40kg/m2
5. Is undergoing active anticoagulant therapy for Deep VeinThrombosis or other conditions (e.g., warfarin, Q10 inhibitors or low molecular weight heparin) or has a history of Deep Vein Thrombosis within the last 6 months or hypercoagulable state.
6. Has had prior venous procedures in the study limb within the last 30 days (including but not limited to, thrombolysis / thrombectomy / stenting / ablation / phlebectomy / sclerotherapy)
7. Has undergone or is expected to undergo any major surgery within 30 days prior to or within 90 days following the study procedure
8. Has a condition, judged by the treating physician, that may jeopardize the patient's well-being and/or confound the results or the soundness of the study
9. Is pregnant or lactating at the time of the study procedure or is intending on becoming pregnant within 90 days following the study procedure
10. Is participating in another clinical study that is contraindicative to the treatment or outcomes of this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Midwest Institute for Minimally Invasive Therapies, Melrose Park, Illinois
  - Vein Clinics of America, Orland Park, Illinois
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - NYU Langone Medical Center, New York, New York
  - UPMC, Pittsburgh, Pennsylvania
  - The Vein Center of Virginia, Norfolk, Virginia
  - Lake Washington Vascular, Bellevue, Washington

REFERENCES:
- [Derived] Gibson K, Elias S, Adelman M, Hager ES, Dexter DJ, Vayuvegula S, Chopra P, Kabnick LS. A prospective safety and effectiveness study using endovenous laser ablation with a 400-mum optical fiber for the treatment of pathologic perforator veins in patients with advanced venous disease (SeCure trial). J Vasc Surg Venous Lymphat Disord. 2020 Sep;8(5):805-813. doi: 10.1016/j.jvsv.2020.01.014. Epub 2020 Mar 21. PMID 32205128

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Veins
Period: Overall Study
Arm/Group | VenaCure EVLT 400 µm Fiber Procedure Kit
Started (Enrolled Population) | 112; 146 Veins
Completed | 70; 113 Veins
Not Completed | 42; 33 Veins

BASELINE CHARACTERISTICS:
Population: ITT Population
Arm/Group | VenaCure EVLT 400 µm Fiber Procedure Kit
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 73
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (5)

OUTCOME MEASURES:

1. Primary Outcome: Acute Primary Ablation Success
Description: The primary effectiveness endpoint is "Acute Primary Ablation Success" defined as complete lack of flow or IPV disappearance in the entire treated segment. Success will be measured via Duplex Ultrasound imaging performed 10 days (± 3 days) post procedure. Primary ablation success must be measured by a physician other than the physician that performed the study procedure.
Time Frame: 10 day
Population: Intent to Treat (ITT) Population
Measure: Count of Units; unit: Veins
Units Other Than Participants: Veins
Arm/Group | VenaCure EVLT 400 µm Fiber Procedure Kit
Number analyzed (Participants) | 83
Number analyzed (Veins) | 125
Veins | 96

2. Secondary Outcome: Technical Success
Description: Technical Success, defined as successful access and entry into the IPV to be ablated and the ability to deliver the intended laser energy, will be evaluated as a secondary endpoint for inclusion in device labeling.
Time Frame: Treatment
Population: Intent to Treat (ITT) Population
Measure: Count of Units; unit: Veins
Units Other Than Participants: Veins
Arm/Group | VenaCure EVLT 400 µm Fiber Procedure Kit
Number analyzed (Participants) | 83
Number analyzed (Veins) | 125
Veins | 119

ADVERSE EVENTS:
Time Frame: 12 months
Description: The safety population was used for all adverse event reporting and analyses.
Groups:
- VenaCure EVLT 400 µm Fiber Procedure Kit (Safety Population): Only one limb can be treated and included in this study; however, multiple IPV's within the study limb may be treated. All IPV's treated will be followed according to the study schedule.
  VenaCure EVLT 400 µm fiber Procedure Kit: The study intervention will be conducted according to the DFU included with the VenaCure EVLT 400 µm fiber Procedure Kit.
Arm/Group | VenaCure EVLT 400 µm Fiber Procedure Kit (Safety Population)
All-Cause Mortality (participants affected / at risk) | 1/93
Serious Adverse Events (participants affected / at risk) | 9/93
Other Adverse Events (participants affected / at risk) | 26/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VenaCure EVLT 400 µm Fiber Procedure Kit (Safety Population) (N=93)
Abscess limb (Infections and infestations) | 1 (1)
Immune thrombocytopenic purpura (Immune system disorders) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Vascular disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Craniocerebral injury (Nervous system disorders) | 1 (1)
Septic shock (Vascular disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VenaCure EVLT 400 µm Fiber Procedure Kit (Safety Population) (N=93)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Procedural pain (General disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Angiodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin injury (Skin and subcutaneous tissue disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Arterial restenosis (Vascular disorders) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Skin ulcer (Vascular disorders) | 3 (3)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02215369/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT02215369/SAP_001.pdf